# Efficacy of Psychological Intervention for Children with Cancer in PIMS Islamabad: A Randomized Controlled Trial

#### Dr. Muhammad Wasim Khan

## **Background:**

Children with cancer and their families experience various psychosocial challenges during and after treatment, including physical and cognitive changes due to medical treatment, alterations in social and familial roles, and the potential threat of death. While most children and families cope and adjust well to the diagnosis and treatment of cancer, a subset of children is at increased risk for anxiety, depression, educational, and relationship difficulties. Caregivers and siblings of pediatric patients are also at risk for heightened distress and post-traumatic stress. Psychosocial care and interventions can play an important role in supporting the well-being of the entire family, beginning at diagnosis.

The psychological impact of cancer on Pakistani children is diverse and far-reaching, ranging from concerns about their future to worries about appearing different from their peers. Given the high prevalence of psychological difficulties among pediatric cancer patients in Pakistan, it is essential to determine the effectiveness of interventions offered to support their mental health and well-being. Studies on cancer patients related to their psychiatric problems are already rare in Pakistan.

## **Objective:**

The main objective of this study is to compare the effect of psychological intervention, such as cognitive-behavioral therapy (CBT), to the routine care given among pediatric oncology patients. The findings of this study will provide evidence to support the integration of psychological intervention strategies into pediatric oncology practice, thus adding new knowledge to the literature and helping improve the care of children with malignancies receiving chemotherapy.

# **Study Design:**

The study will be conducted at the Pediatric Oncology Unit, PIMS, Islamabad. This study will be a two-armed longitudinal, randomized control trial expected to run for six months. Children with malignancy receiving chemotherapy will be recruited and randomly assigned to experimental or control groups.

#### **Intervention:**

The experimental group will receive five sessions of cognitive-behavioral intervention, where maladaptive thoughts and behavior will be identified, behavioral activation will be encouraged, and deep breathing exercises will be practiced. The control group will receive the usual care.

# **Recruitment and Sample:**

The recruitment process will involve the random selection of children diagnosed with malignancies and undergoing treatment at the Pediatric Oncology Unit, the Children's Hospital PIMS Islamabad, Pakistan.

## **Outcome Measures:**

The outcomes will be measured at baseline, post-intervention, and one month after the intervention using the Revised Child Anxiety and Depression Scale and Pediatric Quality of Life Inventory Generic Core Score 4.0.

## **Data Analysis:**

Data analysis will be conducted using SPSS version 23.

## **Ethical Considerations:**

Permission to conduct the study will be acquired from the Ethical Review Board (ERB) of PIMS Islamabad.